CLINICAL TRIAL: NCT01913704
Title: A Randomised Controlled Double Blind Pilot Study Comparing NatroxTM Topical Oxygen Therapy to A Placebo in the Management of Non-Healing Leg Ulcers in Conjunction With Standard Best Practice
Brief Title: Pilot Study Comparing NatroxTM Topical Oxygen Therapy to A Placebo in the Management of Non-Healing Leg Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company turnover
Sponsor: Inotec AMD Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WMC16/CZ/12
Record Dates: First submitted 2013-01-28; First posted 2013-08-01 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Skin Ulcer Venous Stasis Chronic; Mixed Arteriovenous Leg Ulcer
Keywords: venous leg ulcer; mixed aetiology leg ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo device (Placebo Comparator): The placebo comparator is a placebo version of the active device which is a system to deliver oxygen from an oxygen generator topically to the wound bed via a proprietary device.
  The device will be applied to the wound and attached to the placebo oxygen generator and the generator switched on at the time of enrolment. Secondary dressings will then be applied. The device will be removed and reapplied at each dressing change for a treatment period of 6 weeks.
  Interventions: Device: NatroxTM Device
- NatroxTM Device (Active Comparator): A system to deliver oxygen from an oxygen generator topically to the wound via a proprietary device.
  The NatroxTM oxygen delivery device will be applied to the wound and attached to the NatroxTM oxygen generator which will be switched on at the time of first dressing application at enrolment. Secondary dressings will then be applied. The device will be removed and reapplied at each dressing change for a treatment period of 6 weeks.
  Interventions: Device: NatroxTM Device

INTERVENTIONS:
Device: NatroxTM Device — The NatroxTM device is a system to deliver oxygen from an oxygen generator topically to the wound via a proprietary device.
  The NatroxTM ODS oxygen delivery device will be applied to the wound and attached to the oxygen generator and switched on at the time of first dressing application at enrolment. Secondary dressings will then be applied. The oxygen delivery device will be removed and reapplied at each dressing change for a treatment period of 6 weeks.
  Other Names: NatroxTM ODS; NatroxTM Oxygen Generator

SUMMARY:
The purpose of this study is to determine the effectiveness of the NatroxTM Topical Oxygen device versus a placebo in patients with non-healing leg ulceration in conjunction with standard best practice.

DETAILED DESCRIPTION:
Patients will be screened for two weeks before enrollment to assess whether their ulcers are "non-healing", defined as a reduction in wound surface of < 25% after two weeks of standard best practice wound care . On enrolment and randomisation to active or placebo treatment the patient will be treated for six weeks or until 100% epithelialisation, whichever is the sooner, and then treatment will revert to standard best practice, defined as moist wound healing plus compression where appropriate. The reference ulcer will be followed up at two weeks and then at six weeks after the end of the active treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with superficial venous and mixed aetiology leg ulcers on a flat plane in surface area between 4-50cm2
* Patients with diabetes may be included providing they have good metabolic control
* Patients who understand the trial, agree to adhere to the treatment and are able to give consent
* Patients who can be followed by the same investigating team for the whole period of their participation in the study

Exclusion Criteria:

* Patients who present with wounds which are clinically infected and require antimicrobial therapy. Patients who have been treated for a wound infection with antimicrobial therapy (systematically or topically) may be included providing the wound is no longer assessed as infected and there is a two week wash-out period after the last treatment before the patient is reassessed against the inclusion and exclusion criteria
* Patients with a known sensitivity to any of the components of the evaluation device
* Patients with known or suspected malignancy in the wound or surrounding tissue
* Patients whose wounds show a percentage decrease in surface area of >25% during the two week screening period
* Patients who do not have the physical or mental capacity, or a significant other with the ability to change the NatroxTM battery pack on a daily basis
* Patients who present with more than 10% of the wound surface area covered in hard eschar
* Patients who are actively treated with immunosuppressive or cortico-steroidal medication
* Patients who are participating in another clinical trial
* Patients with a known history or poor compliance with medical treatment
* Patients who have been in this trial previously and have withdrawn
* Patients who are unable to understand the aims of the trial and do not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the NatroxTM Topical Oxygen Device | Baseline at week 0 and then at 6 and 12 weeks
  Effectiveness of the NatroxTM Topical Oxygen Device will be established vs. Placebo in patients with non-healing leg ulceration in conjunction with best practice. Effectiveness will measured by the absolute and relative change in wound surface area as measured by digital photography and wound-mapping software.

SECONDARY OUTCOMES:
Change in the wound pain over the study duration | Baseline at week 0, and then each weekly dressing change, 8 weeks and 12 weeks
  Measured using a validated Visual Analogue Scale ranging from 0 to 10
Patient comfort with the device at dressing change | first removal of device and then on subsequent weekly changes
  Patient will be recorded on each visit with the dressing applied and will be recorded as a yes/no to comfort experienced by the patients
Patient acceptability of the device during wear | Each weekly dressing change until week 6
  Patient questioned as to ability to mobilise, comfort of dressing and device and possible disturbance of sleep patterns, answers recorded as yes/no
Statistical information from which to power a future large multi-centre randomised trial | Study End at week 12
  Statistical information on use of Natrox device and effectiveness on patients. Wound surface area will be measured in square centimetres as defined by wound mapping software. The wound surface area reduction between six weeks and baseline will then be calculated. Wound surface area will be measured at weekly intervals for the 6 weeks of active treatment and then at weeks 8 and 12 for follow up. The primary analysis will be an intent-to-treat analysis. A two-sided significance level of 0.05 will be used for all analyses. A general linear model taking into account the treatment groups and centres (surgical and dermatology clinics) as fixed effects and a baseline wound surface area as a covariate will be used to test the null hypothesis of similar effects in surface area reduction between treatment groups.
Efficiency of Exudate transportation through the device to the secondary dressing | weekly up to week 6 (end of natrox treatment period)
  Measured by the frequency of changes of the secondary dressing and by recording the incidence of maceration.
Improvement in the wound bed during treatment with Natrox and Oxygen Delivery System (ODS) | Baseline at week zero, weekly and end of treatment at week 6
  Measured by visual assessment weekly by the Investigators
Reliability of the protocol | Study end follow up at week 12
  The reliability of the protocol will be determined by ability to implement it in the clinical setting effectively and the accuracy of the outcomes delivered from the study
Monitor the safety of the device in use | Study treatment end at week 6 and then until follow up at 12 weeks
  Measured by recording the incidence and severity of adverse events as reported.

CONTACTS AND LOCATIONS:
Overall Officials: R Gurlich, Professor, Principal Investigator — Fakultni Nemocnice Kralovske Vinohrady Prague
Locations (2):
- Czechia (2):
  - Fakultni Nemocnice Kralovske Vinohrady, Clinical of Surgery, Prague
  - Fakultni Nemocnice Kralovkse Vinohrady, Clinic of Dermatology, Prague